CLINICAL TRIAL: NCT06984900
Title: Investigating The Effect of Short-Term Aerobic Exercise on Stress and Mood Among Students
Brief Title: How Short-Term Aerobic Exercise Affects Stress and Mood in Students
Acronym: SEAEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Feras Alsultan, Principal Investigator (PI), Qassim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-71-12
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Mental Health; Well-Being; Exercise; Stress; Mood
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short-Term Aerobic Exercise Group (Experimental)
  Interventions: Other: Group Aerobic Exercise Session

INTERVENTIONS:
Other: Group Aerobic Exercise Session — The Aerobic Exercise Program is designed to improve mood and reduce stress among university students through structured, moderate-intensity aerobic activities.
  Session Structure: Participants engage in moderate-intensity aerobic exercises such as treadmill walking or running, tailored to individual fitness levels, ensuring accessibility and inclusivity. Each session consists of a 10-minute warm-up, 30 minutes of aerobic exercise, and a 5-minute cool-down.
  This intervention incorporates a dual assessment approach using the Profile of Mood States (POMS) and the Perceived Stress Scale (PSS) to evaluate mood and stress levels both before and after exercise. Participants complete these assessments multiple times, allowing for a nuanced understanding of how aerobic exercise influences mood and stress over time.

SUMMARY:
This study was conducted to understand how short-term aerobic exercise affects mood and stress in university students. The research focused on healthy male and female students between the ages of 18 and 25. Participants were asked to complete two questionnaires: one to measure their mood and another to assess their stress levels. These questionnaires were filled out before, immediately after, and at several intervals up to 24 hours after a single session of aerobic exercise.The goal was to see whether exercise could quickly improve mood and reduce stress, and how long these effects might last. The study was carefully designed, and ethically approved. By focusing on immediate and short-term changes, the research highlights the potential benefits of exercise for mental well-being in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female students aged between 18 and 25 years.
* Ability to speak and understand written English.

Exclusion Criteria:

* Students who are pregnant or planning to become pregnant.
* Students who currently smoke.
* Students who respond "yes" to any of the seven questions on the Physical Activity Readiness Questionnaire (PAR-Q).
* Students taking medications for chronic diseases such as high blood pressure or diabetes.
* Students with a current or past diagnosis of a psychotic disorder.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Total Mood Disturbance Following Short-Term Aerobic Exercise in University Students | TMD is assessed at eight time points: Before exercise (T0) Immediately after exercise (T1) At intervals: 1 hour (T2), 2 hours (T3), 4 hours (T4), 8 hours (T5), 12 hours (T6), and 24 hours post-exercise (T7).
  Total Mood Disturbance (TMD):
  Measured using the Profile of Mood States (POMS) questionnaire.
  Scores range from 0 to a maximum depending on the number of items (65 items rated on a 0-4 Likert scale, resulting in a theoretical range of 0 to 260).
  A higher TMD score represents a worse overall mood outcome.
Perceived Stress Levels Following Short-Term Aerobic Exercise in University Students | Assessed at two time points: Before exercise (T0) 24 hours after exercise (T7).
  Perceived Stress Levels:
  Measured using the Perceived Stress Scale (PSS). Scores range from 0 to 40.
  Higher scores indicate higher levels of perceived stress. Scores can be categorized as:
  Low stress: 0-13 Moderate stress: 14-26 High stress: 27-40

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University, in Qassim University Medical City, the Kingdom of Saudi Arabia (KSA)., Buraidah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The study aims to share individual participant data (IPD) with other researchers for further analysis and to enhance the understanding of the effects of aerobic exercise on mood and stress among students.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be made available upon request. Requests can be submitted to the principal investigator.